



## **ADOLESCENT ASSENT FORM FOR YOUTH AGES 12-17**

Nemours Template January 2024

Your parent has given permission for you to be in a project called a research study. But first, we want to tell you all about it so you can decide if you want to be in it. If you don't understand, please ask questions. You can choose to be in the study, not be in the study or take more time to decide.

# 1. What is the name of the study?

Using Ultrasound as an Alternative to Radiography in Measuring Magnetically Controlled Growing Rods (MCGR) in Tibia and Femur Lengthening Patients

## 2. Who is in charge of the study?

The doctor in charge of the study is Dr. Jason Malone

### 3. What is the study about?

We would like to find out if ultrasound imaging is a viable alternative to x-rays in assessing bone lengthening measurements.

## 4. Why are you asking me to be in this study?

You are being asked to be in the study because you are a pediatric patient at Nemours undergoing a tibia or femur lengthening procedure with an intramedullary mechanical rod.

#### 5. What will happen to me in the study?

- All patients will follow up weekly for clinical exam and imaging with no change to standard of care.
- All patients will obtain standard AP and Lateral x-rays
- All enrolled patients will have ultrasound imaging and measurements in the same locations as the x-rays.
- All measurements will be stored in a password protected file with no patient identifiers and will be safely discarded at the end of the study.

#### 6. Will I be paid to be in this study?

You will not be paid for being in this study.

## 8. Do I have to be in the study?

You don't have to do the study if you don't want to. If you are in the study, you can stop being in it at any time. Nobody will be upset with you if you don't want to be in the study or if you want to stop being in the study. The doctors and nurses will take care of you as they have in the past. If you have any questions or don't like what is happening, please tell the doctor or nurse.

You have had the study explained to you. You have been given a chance to ask questions. By writing your name below, you are saying that you want to be in the study.





| Name of Adolescent ( <b>Print</b> ) | |
|--------------------------------------------------|------|
| Signature of Adolescent | Date |
| Name of Person Obtaining Assent ( <b>Print</b> ) | |
| Signature of Person Obtaining Assent | Date |

Nemours Template January 2024